CLINICAL TRIAL: NCT05659693
Title: The Effect of Digital Literacy Education Given to Postmenopausal Women on Health Literacy and Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Selcan Bakır, Clinical Nurse, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-74555795-050.01.04-519850
Record Dates: First submitted 2022-11-30; First posted 2022-12-21 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Postmenopausal Symptoms; Literacy; Quality of Life; Health Literacy; Digitalism
Keywords: Postmenopausal Symptoms; digital literacy; Quality of Life; Health Literacy; menopause
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Intervention Model Description: Type of Study: This study is a randomized controlled trial. The pre-test-post-test will be carried out with a pattern.
Who Masked: Participant, Investigator
Masking Description: Women who meet the inclusion criteria will be included in the sample using a simple random method. Before the research numbers were produced from random.org, envelopes of the same size and characteristics were created for each participant by a person other than the researcher (IU-C, Research Assistant B.Y) and numbers between 1 and 120 were written on them. Then, considering the data losses, numbers from 1 to 120 were generated from random.org. The researcher will use online "spinning games" (https://www.kodvizit.com/cekilis/cark) while dividing the participants into groups. Numbers from 1-120 will be written on the online wheel on the site. The researcher will first apply a digital literacy scale to the woman who accepts the research. The woman with a scale score of 3.40 and below will be asked to spin the wheel from the online "spinning games" site and the experimental - control group will be determined.
  Experimental Group: 50 people Control Group: 50 people
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Digital literacy education specific to menopause will be given to this group.
  Interventions: Behavioral: digital literacy education specific to menopause
- Control Group (No Intervention): no intervention will be applied to this group.

INTERVENTIONS:
Behavioral: digital literacy education specific to menopause — Education; It is planned as 5 sessions in the form of presentation, homework, scenario and sending reminder messages. The training is planned to last approximately 20 minutes with a power point presentation prepared by the trainer. The survey will be evaluated in the first session. Women will be told what digital literacy is, why it is important, how to verify information and resources, security of accounts, resources, money and devices, access to information, understanding and valuing information. A screening and access to information session will be held with a scenario prepared on menopausal symptoms, taking into account the variables of information and resource security, access to information, understanding and valuing information, with examples on the digital platform. The woman will be given a scenario homework on menopausal symptoms. Interim evaluation will be made in the fourth week of the training. The final evaluation will be made in the fifth session.
  Arms: Experimental Group

SUMMARY:
During menopause, women may experience many conditions and symptoms due to fluctuation in hormone levels. These symptoms can affect a woman's social and personal functioning and quality of life. The symptoms and quality of life experienced by women during menopause are closely related to health literacy and digital literacy levels.

Women in the menopausal period often turn to alternative and complementary practices to cope with the symptoms. They obtain this information from Web 2.0 technologies (Instagram, Facebook, etc.) and other sources on the internet, along with the innovations brought by the developing world. However, they do not have enough skills to question the reliability and accuracy of the information sources they obtain. In this context, digital literacy emerges as a new concept in today's digital transformation. Digital Literacy is the awareness, attitude and ability of individuals to use digital tools and possibilities appropriately to identify, access, manage, integrate, evaluate, analyze and synthesize digital resources, create new information, create media expressions and communicate with others. With the developing technology and widespread use of the internet, the impact of the information obtained from digital platforms on the current health literacy and quality of life of women is gaining importance.

In the literature, it has been determined that the relationship between digital literacy, health literacy and quality of life has been examined in different samples such as the elderly and individuals with chronic diseases. However, no research has been found in the literature examining the effect of a planned digital literacy education specific to menopause on the health literacy and quality of life of postmenopausal women.

The age group in which the research is planned is a group that can use Web 2.0 technologies (Instagram, Facebook, etc.) and other sources on the internet, but we think that they have limited information about accessing information sources and examining the accuracy of the information they have obtained. In this context, we believe that a planned digital literacy education specific to menopause will increase the health literacy and quality of life of postmenopausal women.

DETAILED DESCRIPTION:
Purpose of the Study: This study was planned as a randomized controlled experimental study to examine the effect of digital literacy education given to postmenopausal women on health literacy and quality of life.

Data Collection: The data will be collected by the researcher by face-to-face interview method in a total of 5 sessions, each session of 30 minutes.

Statistical Methods to be Used: SPSS program will be used in the analysis of the obtained data. The conformity of the data to the normal distribution will be examined by considering the Shapiro-Wilk test; Parametric methods will be used in the analysis of normally distributed variables, and non-parametric methods will be used in the analysis of non-normally distributed variables. Independent-Samples T test, Mann-Whitney U (Exact) test and T test for Dependent Groups, Wilcoxon test will be used in the comparison of 2 independent groups. PearsonCorrelation, Spearman'srho tests will be used to examine the correlations of the variables with each other. Comparison of categorical data will be tested with PearsonChi-Square and FisherExact tests.

ELIGIBILITY:
Inclusion Criteria:

* Being between 45 - 65 years old,
* Being in the postmenopausal period
* Using a smart phone, tablet and/or computer
* Digital literacy level of 3.40 and below

Exclusion Criteria:

* Having a diagnosed psychiatric disorder
* Having a diagnosed cancer disease

  * Scale item total score is in the high range between 3.41-4.20 and very high between 4.21-5.00 (Ng, 2012).

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
digital literacy education increases the digital literacy level of women | The change in the digital literacy scale score of the participants in 2 months was evaluated with the digital literacy scale. Participants were expected to have an increase in their scores during this time.
  Digital Literacy Scale: The Digital Literacy Scale (DFLS) developed by Ng (2012) consists of 17 items. The scale items are answered by the participants in a 5-point Likert structure as "5: Strongly agree, 4: Agree, 3: Undecided, 2: Disagree, 1: Strongly disagree". The lowest score that can be obtained for the whole scale is 17 and the highest score is 85. While interpreting the mean score of the scale; Score ranges were used between 1.00-1.80 very low, 1.81-2.60 low, 2.61-3.40 medium, 3.41-4.20 high, 4.21-5.00 very high. Low scores from the overall Digital Literacy scale indicate low Digital Literacy level, while higher scores indicate high digital literacy.
digital literacy education increases women's health literacy level | The change in the health literacy scale score of the participants in 2 months was evaluated with the health literacy scale. Participants were expected to have an increase in their scores during this time.
  Health Literacy Scale: It is the scale of the 47-item HealthLiteracySurvey in Europe (HLS-EU) form developed by Sorensen (2012) and later simplified by working together again by Toçi, Bruzari and Sorensen. The Health Literacy scale consists of 25 items and four sub-dimensions. The lowest score for the whole scale is 25 and the highest score is 125. The items in the scale are answered by the participants in a 5-point Likert structure as "5: I have no difficulty, 4: I have little difficulty, 3: I have a little difficulty, 2: I have a lot of difficulty, 1: I am unable to do / I have no ability / impossible". Low scores indicate that the Health Literacy status is insufficient, problematic and weak, while high scores indicate that it is sufficient and very good. As the score obtained from the scale increases, the health literacy level of the individual increases.
digital literacy education improves women's menopause-specific quality of life | The change in the participants' menopausal symptoms and coping skills at 2 months was evaluated with The Menopause-Specific Quality of Life Questionnaire. Participants were expected to have an increase in their scores during this time.
  The Menopause-Specific Quality of Life Questionnaire (MENQOL) was developed by Hilditch et al. in 1996 in order to evaluate the quality of life of menopausal women. The scale consists of 29 Likert type questions and 4 sub-domains: vasomotor (questions 1-3), psychosocial (questions 4-10), physical (questions 11-26) and sexual (questions 27-29). The score for each question ranges from 1 to 8. In the scoring, 1 point indicates that the situation did not occur, 2 points indicate that the situation did occur, but it was not disturbing, and a score between 3-8 indicates the severity of the situation. High scores on the scale indicate low quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: selcan bakır, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- İstanbul university -cerrahpaşa, faculty of nursing, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The information obtained from this study will be used for research purposes and personal information will be kept confidential; however, the data may be used for publication purposes. 2 years after the completion of the study, the data will be destroyed by the destruction machine belonging to the institution and will be kept locked in a closed cabinet during this period.